CLINICAL TRIAL: NCT07071779
Title: Web-based Alcohol-specific Inhibition Training in Adolescents and Young Adults With Alcohol Use Disorder
Acronym: WAIT-AYA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: BASEC2024-01150
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Alcohol Use Disorder (AUD)
Keywords: Alcohol use disorder; Alcohol-specific inhibition training; Cognitive bias modification; Feasibility pilot randomized controlled trial
MeSH Terms: conditions — Alcoholism | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alcohol-specific inhibition training (Experimental): 12 sessions of alcohol-specific inhibition training
  Interventions: Other: Alcohol-specific inhibition training
- Control training (Active Comparator): 12 sessions of unspecific inhibition training
  Interventions: Other: Control training

INTERVENTIONS:
Other: Alcohol-specific inhibition training — Twelve sessions of alcohol-specific inhibition training
  Arms: Alcohol-specific inhibition training
Other: Control training — Twelve sessions of unspecific inhibition training
  Arms: Control training

SUMMARY:
Alcohol misuse is one of the most common risk factors for health problems and premature death among adolescents and young adults worldwide. Although there are effective treatments for alcohol use disorder (AUD), there is still a need to further improve their effectiveness and make them easier to access. Early research suggests that alcohol-specific inhibition training, when used in addition to specialized treatment, can improve treatment outcomes. This training aims to strengthen inhibition specifically in situations related to alcohol. The goal of this project is to offer this training for the first time in the form of a smartphone app, which is expected to increase the availability of the training. The main aim of the study is to evaluate whether this new app-based cognitive training is feasible as an add-on to the treatment of AUD in adolescents and young adults. In addition, the study will gather initial insights into whether the training affects drinking behavior and related brain processes. The project will be conducted as a double-blind, clinical pilot study. A total of 210 adolescents and young adults between 14 and 27 years old will be recruited from five specialized treatment centers. After the first study visit, participants will be randomly assigned to one of two groups: (1) an intervention group receiving the alcohol-specific inhibition training or (2) a control group receiving a similar alcohol-nonspecific inhibition training. During their participation, all participants will complete six short training sessions with the app. About one month later, they will complete six additional booster training sessions. This research may help develop effective, easily accessible tools to support young people with alcohol use disorder.

ELIGIBILITY:
Inclusion Criteria:

* Age 14 - 27 years
* Alcohol use disorder identification test (AUDIT) ≥ 8
* Alcohol use disorder scale (AUD-S) ≥ 2
* Currently undergoing outpatient treatment or online counselling in one of 5 specialized treatment settings
* Sufficient German language skills
* Informed Consent as documented by signature
* Owner of a smartphone with internet access

Exclusion Criteria:

* Other severe substance use (except nicotine and cannabis) determined by the cut-off value ≥ 25 in the drug use disorder identification test (DUDIT)
* Current medical conditions excluding participation
* Inability to read and understand the participant's information
* Enrolment of the investigator, his/her family members, employees, and other dependent persons

Additional exclusion criteria for Electroencephalography (EEG)-substudy:

* Current medication affecting EEG (e.g., benzodiazepines)
* Other severe substance use determined by the cut-off value ≥ 25 in the DUDIT (except nicotine)
* History of epilepsy

Ages: 14 Years to 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants recruited | From enrollment to the last assessment, approx. 16 weeks
  Number of participants recruited during the recruitment period in all participating clinical centers is one indicator of the feasibility of implementing alcohol-specific inhibition training in a smartphone app.
Number of participants successfully completing the program | At the last assessment, approx. 16 weeks from enrollment
  Number of participants successfully completing the program is one indicator of the feasibility of implementing alcohol-specific inhibition training in a smartphone app.
Proportion of participants completing the follow-up visits | At the last assessment, approx. 16 weeks from enrolment
  Proportion of participants completing the follow-up visits is another indicator of feasibility.
Number of participants adhering to the treatment | From enrollment to last last training session, approx. 10 weeks
  Number of participants adhering to the treatment, i.e. participating in all planned twelve training sessions, is another indicator of feasibility of implementing alcohol-specific inhibition training in a smartphone app.
Number of adverse events | From enrollment to the last assessment, approx. 16 weeks
  Number of adverse events is another indicator of feasibility of implementing alcohol-specific inhibition training in a smartphone app.

SECONDARY OUTCOMES:
Percentage of days abstinent | At the last assessment, approx. 16 weeks from enrolment
  Percentage of days abstinent is the main secondary outcome indicating preliminary effects on drinking behavior. It is measured by the Timeline Follow-Back method at 3-month follow-up.
Number of heavy drinking days | At the last assessment, approx. 16 weeks from enrolment
  Number of heavy drinking days is another secondary outcome indicating preliminary effects on drinking behavior. It is measured by the Timeline Follow-Back method at 3-month follow-up.
P3-component of event-related potentials | 4-6 weeks.
  The P3-component of event-related potentials measured with electroencephalography (EEG) is used as a secondary outcome in the EEG- substudy to investigate whether iAlc-IT modifies the neurophysiology of alcohol-specific inhibition
N2-component of event-related potentials | 4-6 weeks.
  The N2-component of event-related potentials measured with electroencephalography (EEG) is used as a secondary outcome in the EEG- substudy to investigate whether iAlc-IT modifies the neurophysiology of alcohol-specific inhibition

CONTACTS AND LOCATIONS:
Overall Officials: Maria Stein, PD Dr., Principal Investigator — University of Bern
Locations (1):
- University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
The decision to share IPD depends on the explicit consent provided by participants as part of the informed consent process. Since it is not possible to determine in advance whether participants will grant permission for data sharing, IPD sharing is not planned.